CLINICAL TRIAL: NCT00385879
Title: The Effects of Case Management in a Medicaid Managed Care Plan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Metropolitan Jewish Health System (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Health Plus at Home
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-10

CONDITIONS: Neoplasms; Heart Diseases; Adrenal Cortex Diseases
MeSH Terms: conditions — Neoplasms; Heart Diseases; Adrenal Cortex Diseases | interventions — Case Management

INTERVENTIONS:
Behavioral: Case management

SUMMARY:
The purpose of this study is to evaluate whether or not case management by a social worker and nurse can decrease the number of emergency room visits, increase the number of primary care doctor visits, and increase quality of life of people in a Medicaid managed care plan.

DETAILED DESCRIPTION:
This study will assign participants based on Zip Code to one of two conditions: control and experimental. In the control group, participants will receive telephonic assessments at baseline, three months, and six months. These assessments will be conducted by a member of the Medical Center's Department of Geriatrics under the supervision of the Principal Investigator. Participants in the experimental group will receive medical case management provided by a nurse and social worker in the homecare setting including an in-home assessment. Assessments will be conducted at baseline, three months, and six months during routine homecare visits. Dependent variables being measured include: access to primary care physicians, emergent hospitalizations/admissions, articulation of advance directives, and quality of life. Data will be collected through the participants' medical claims and records to analyze the number of emergent hospitalizations/admissions, documentation of advance directives, and number of visits to primary care physicians. To measure participants' quality of life, the Depression Self-Rating Scale and the Clinical Anxiety Scale will be utilized. Data will be compared between and within the groups via statistical analyses. The researcher will conduct pre-post comparisons of utilization and other database-derived outcomes for both groups, comparing the 12 months prior to and up to 20 months following enrollment.

ELIGIBILITY:
Inclusion Criteria:

* participation in a Medicaid managed care plan
* resident of identified zip codes in Brooklyn, NY
* frequent hospitalizations and low frequency of primary doctor visits

Exclusion Criteria:

* residents outside the catchment area
* patients not being managed in a Medicaid managed care plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2006-05; Study Completion 2008-01

PRIMARY OUTCOMES:
The outcome measure for the number of emergency room visits will be calculated from the medical record counting the number of hospital emergency room visits; for access to primary physicians, the medical record will be reviewed as well.

SECONDARY OUTCOMES:
The outcomes for quality of life will be evaluated from the McGill Quality of Life Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Paris, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Metropolitan Jewish Health System, Brooklyn, New York, United States

REFERENCES:
- [Result] Chattopadhyay A, Bindman AB. The contribution of Medicaid managed care to the increasing undercount of Medicaid beneficiaries in the Current Population Survey. Med Care. 2006 Sep;44(9):822-6. doi: 10.1097/01.mlr.0000218835.78953.53. PMID 16932133